CLINICAL TRIAL: NCT03032744
Title: Aligning With Schools To Help Manage Asthma
Brief Title: Aligning With Schools To Help Manage Asthma (Project ASTHMA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Lucy Holmes, MD, Clinical Associate Professor of Pediatrics, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IMPACT1; UL1TR001412 (NIH)
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Asthma
Keywords: Pediatric; School Based Health Center
MeSH Terms: conditions — Asthma | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Intervention group will receive the morning dose of their daily preventive asthma medication at school. The student & family will be responsible to administer the evening dose & both doses on non-school days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): All participants will undergo an initial asthma assessment per the NAEPP-EPR3 (National Asthma Education and Prevention Program - Expert Panel Report 3) guidelines, as well as asthma education. Participants randomized to the intervention group will be prescribed the appropriate asthma therapy based on their assessment (i.e. providing 'asthma assessment & management'), and receive the morning dose of their daily asthma controller medication at school on school days.
  Interventions: Other: Asthma Assessment & Management; Other: Asthma Education; Other: Controller medication at school
- Usual Care (Active Comparator): All participants will undergo an initial asthma assessment per the NAEPP-EPR3 (National Asthma Education and Prevention Program - Expert Panel Report 3) guidelines, as well as asthma education. Participants randomized to the usual care group will be provided with the results of their asthma assessment and be instructed to follow up with their primary care provider. They will continue to receive all of their daily asthma controller medication at home.
  Interventions: Other: Asthma Assessment & Management; Other: Asthma Education

INTERVENTIONS:
Other: Asthma Assessment & Management — Asthma Assessment & Management based on NAEPP-EPR3 guidelines
Other: Asthma Education — Asthma education on medications
Other: Controller medication at school — Students will receive the morning dose of their daily preventive asthma medication at school on school days.
  Arms: Intervention

SUMMARY:
Project ASTHMA is a school-based health center intervention program that institutes guideline-based chronic asthma care and provides supervised administration with daily preventive asthma medications to improve asthma symptoms and lung function, reduce emergency visits, and decrease missed days of school among children from communities with health disparities.

DETAILED DESCRIPTION:
Project ASTHMA in schools is a 7 month randomized control intervention pilot trial. Forty students, ages 4 to 14 years, with persistent asthma, or who utilize acute care facilities frequently for their asthma, will be recruited from 3 urban SBHCs in the fall of 2018. All students will receive NHLBI guideline-based asthma assessments to determine eligibility and proper dosing of preventive medication. The asthma assessment will include spirometry testing. All enrolled students and parents will receive asthma education at the time of enrollment. Eligible students will be randomized to an intervention or usual care group using permuted block randomization stratified by SBHCs. In collaboration with the student's PCP, the SBHCs' mid-level providers will prescribe the preventive medication to the students in the intervention group. These students will receive the morning dose of their preventive medication from the school nurse each school day for the remainder of the school year. Students and their parents will be responsible to administer the evening and non-school day doses. Students randomized to the usual care group will be referred back to their PCP for further asthma management. All participants will be re-evaluated at 1, 3 and 7 months after enrollment, and medication dose adjustments will be made in the intervention group as needed.

ELIGIBILITY:
Inclusion Criteria:

* Active asthma
* Diagnosed with asthma for at least 12 months
* Enrolled in the school-based health center
* Persistent asthma as defined by NAEPP-EPR3 guidelines OR at least 1 hospitalizations OR at least 2 ED/urgent care visits OR at least 2 courses of oral steroids for asthma in the previous 12 months for asthma

Exclusion Criteria:

* Underlying heart or lung disease other than asthma
* Student has well controlled asthma

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucy C Holmes, MD, MPH, Principal Investigator — University at Buffalo
Locations (1):
- John R. Oishei Children's Hospital, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holmes LC, Orom H, Lehman HK, Lampkin S, Halterman JS, Akiki V, Supernault-Sarker AA, Butler SB, Piechowski D, Sorrentino PM, Chen Z, Wilding GE. A pilot school-based health center intervention to improve asthma chronic care in high-poverty schools. J Asthma. 2022 Mar;59(3):523-535. doi: 10.1080/02770903.2020.1864823. Epub 2021 Jan 6. PMID 33322963

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 13 | 16
Completed | 12 | 15
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Continuous [Mean (Full Range); unit: years] | 8.6 [4 to 14] | 9.2 [4 to 14] | 8.9 [4 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 14 | 24
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Asthma Control Test (ACT) [Mean (Standard Deviation); unit: units on a scale] — Asthma Control Test (ACT) ACT test is a screening tool to assess how well controlled a patient's asthma is Minimum: 0 Maximum: 27 Higher scores are better. Scores less than 19 are considered not well controlled asthma
  units on a scale | 14.8 (4.27) | 14.4 (4.96) | 14.6 (4.59)

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Days Per Week, in the Previous 4 Weeks, of Daytime Asthma Symptoms From Baseline to 7-month Follow-up
Description: Total number of days per week, over the previous 4 weeks, of asthma symptoms Minimum: 0 Maximum: 7 Lower number indicates improvement The change in number of days per week of asthma symptoms from baseline to 7-month follow-up
Time Frame: Baseline, 1-month, 3-month, 5-month, 7-month
Measure: Mean (95% Confidence Interval); unit: days per week
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 12 | 15
days per week | -3.4 [-4.9 to -1.9] | -2.8 [-4.1 to -1.2]

2. Secondary Outcome: Change in ACT Score From Baseline to 7-month Follow-up
Description: Improvement in ACT (Asthma Control Test) score, a validated questionnaire for the assessment of asthma symptoms, which is included in the NAEPP-EPR3 guidelines for components of control. Minimum value is 0. Maximum value is 27. Higher scores mean a better outcome. Scores less than 19 suggest not well-controlled asthma.
  The change in ACT score from baseline to 7-month follow-up
Time Frame: Baseline, 1-month, 3-month, 5-month, 7-month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 12 | 15
score on a scale | 6.4 [3.2 to 9.4] | 8.3 [5.1 to 10.8]

3. Secondary Outcome: Change in FEV1/FVC Ratio From Baseline to 7-month Follow-up
Description: Improvement FEV1/FVC ratio on spirometry. Higher number is a better outcome. FEV1/FVC ratio is a calculation used in pulmonary function testing to help diagnose lung conditions, particularly obstructive and restrictive lung diseases. It represents the proportion of air a person can exhale in the first second of a forced expiration (FEV1 - forced expiratory volume in 1 second) compared to the total amount of air they can exhale with maximal effort (FVC - forced vital capacity).
  The change in FEV1/FVC ratio from baseline to 7-month follow-up.
Time Frame: Baseline, 1-month, 3-month, 5-month, 7-month
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 12 | 15
ratio | 0 [-0.01 to 0.04] | -0.05 [-0.07 to -0.02]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/16
Other Adverse Events (participants affected / at risk) | 0/13 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT03032744/Prot_SAP_000.pdf
  • Informed Consent Form: Parent (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT03032744/ICF_001.pdf
  • Informed Consent Form: Assent - 14 years old (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT03032744/ICF_002.pdf
  • Informed Consent Form: Assent - 7-13 yrs old (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT03032744/ICF_003.pdf